CLINICAL TRIAL: NCT04665544
Title: Prospective Observational Study on Sentinel Node Biopsy Using Two Concurrent Labelling Techniques (Radioactive Tracer With/Without Blue Dye vs. Indocyanine Green-ICG) in Early-stage Endometrial Cancer Patients (TESLA-1).
Brief Title: Tracers for Endometrial Cancer Sentinel Node Labeling
Acronym: TESLA-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Maja Pakiz, Dr., University Medical Centre Maribor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEEGOG EX-02
Record Dates: First submitted 2020-11-18; First posted 2020-12-11 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-04

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early-stage endometrial cancer patients (Experimental): * Histologically proven endometrial cancer (any tumour type).
  * Apparent early-stage endometrial cancer with intermediate or high risk prognostic factors (deep myometrial invasion or G2/G3 disease or non- endometrioid histological type), no evidence of bulky or suspicious pelvic/para-aortic lymph nodes or distant metastases on preoperative conventional imaging studies; minimum requirement for clinical staging includes expert US or pelvic MRI for local staging and abdominal US or abdominal CT scan or PET CT for distant staging.
  * Performance status ECOG: 0-1.
  * Age ≥18, ≤85.
  * History of second primary cancer only if more than 5 years with no evidence of disease.
  * Approved and signed informed consent
  Interventions: Procedure: SLN side-specific detection rate using radioactive tracer with/without blue dye and ICG tracer.

INTERVENTIONS:
Procedure: SLN side-specific detection rate using radioactive tracer with/without blue dye and ICG tracer. — The primary objective of this study is to compare SLN detection rate using two types of intracervical tracers (radioactive tracer with or without blue dye vs. ICG).
  The null hypothesis is that the detectionrate does not differ between the two techniques.

SUMMARY:
Sentinel lymph node (SLN) biopsy is currently used in the management of vulvar and breast cancers as well as in malignant melanoma, and is being intensively studied in patients with cervical and endometrial cancers. The role of lymphadenectomy in the surgical management of early-stage endometrial cancer is still controversial. The main reason to perform a SLN biopsy is to detect the lymph node that will be the first involved with metastatic disease in the nodal basin. The SLN biopsy is performed after the SLN is located with the use of different tracers in a concept called SLN mapping. Moreover, SLN evaluation has been reported to improve the accuracy of lymph node staging due to SLN pathologic ultrastaging, which includes multiple serial sectioning and immunohistochemical assessment. The aim of this project is to conduct a multicentre, prospective, observational trial to compare two different SLN labelling methods (radioactive tracer with/without blue dye vs. indocyanine green-ICG) in the same patient and to evaluate the unilateral detection rate, sensitivity, number of detected SLN, anatomical localisation of detected SLN and bilateral detection rate of SLN. The main aim of the trial is the comparison of SLN mapping between two SLN labelling methods in the same patient. The trial will answer a question whether a combination of labelling methods in the same patient increase importantly the sensitivity of SLN biopsy.

The trial has a high potential to reach the calculated number of cases and thus bring in evidence/data that will be essential for future management of SLN biopsies in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven endometrial cancer (any tumour type).
* Apparent early-stage endometrial cancer with intermediate or high risk prognostic factors (deep myometrial invasion or G2/G3 disease or non- endometrioid histological type), no evidence of bulky or suspicious pelvic/para-aortic lymph nodes or distant metastases on preoperative conventional imaging studies; minimum requirement for clinical staging includes expert US or pelvic MRI for local staging and abdominal US or abdominal CT scan or PET CT for distant staging.
* Performance status ECOG: 0-1.
* Age ≥18, ≤85.
* History of second primary cancer only if more than 5 years with no evidence of disease.
* Approved and signed informed consent form to participate in the study.

Exclusion Criteria:

* Pregnancy
* Desire for fertility sparing
* History of pelvic or abdominal radiotherapy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
SLN unilateral detection rate | 2 years
  Number of hemipelvises where the SLN was found/number of all hemipelvises for each tracer and combination of tracers

SECONDARY OUTCOMES:
Sensitivity of SLN biopsy for pelvic lymph node staging. Anatomical localisation of detected SLN | 2 years
  Number of true positive LN/(number of true positive LN+number of false negative LN) for each tracer and combination of tracers
Number of detected SLN. | 2 years
  Average number of detected SLN (in the specimen, labelled with the tracer, there might be one or more LN; the number of removed LN is one of the quality indicator).
Descriptive meassure: Anatomical localisation of detected SLN | 2 years
  Exact anatomical localisation of SLN (1-external iliac vessels, 2-internal iliac vessels, 3-obturator region, 4-paraaortic region, 5-presacral region).
Bilateral detection rate. | 2 years
  The number of patients with bilateral SLN detection/the number of all patients for each tracer and combination of tracers

CONTACTS AND LOCATIONS:
Overall Officials: Maja Pakiž, MD,PhD, Study Chair — University Medical Centre Maribor
Locations (6):
- Czechia (4):
  - University Hospital Ostrava, Ostrava
  - Charles University-First Faculty of Medicine, University Hospital Bulovka, Department of Gynecology and Obstetrics, Prague
  - Gynecologic Oncology Center, Department of Obstetrics and Gynecology; First Faculty of Medicine, Charles University of Prague and General Hospital in Prague, Prague
  - KNTB Zlin, Zlín
- Department of Gynecology, Gynecologic Oncology and Endocrinological Gynecology, Medical University of Gdansk, Gdansk, Poland
- University Medical centre Maribor, Department for Gynecologic and Breast Oncology, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No